CLINICAL TRIAL: NCT01202981
Title: Impact of IOL Glistenings on Visual Quality and Function in Patients Implanted With a Single-Piece AcrySof IOL That Exhibits Glistening Formation
Brief Title: Impact of Glistenings in AcrySof Intraocular Lenses on Visual Quality
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 42093
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Lenses, Intraocular; Glistenings; Visual Quality
Keywords: glistenings; contrast sensitivity; visual quality; straylight; AcrySof IOL

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Patients who had cataract surgery by the Investigators between July 1, 2007 and June 30, 2008.
- Group 2: Patients who had cataract surgery by the Investigators between July 1, 2008 and July 1, 2009.

SUMMARY:
This study will assess the impact of IOL glistenings on visual quality and function in patients implanted with a single-piece AcrySof intraocular lens (IOL) that exhibits glistening formations. The primary objective is to determine if random light scattering (measured by C-Quant)correlates with severity of glistenings, other objective measures of visual function (visual acuity, low contrast visual acuity, low contrast visual acuity with glare), and subjective measures of patients' perceptions of their visual quality after cataract surgery (quality of life survey, reports of symptomology and satisfaction).

ELIGIBILITY:
Inclusion Criteria:

1. Presence of obvious glistenings by slit lamp exam
2. Best spectacle corrected visual acuity of 20/20 or better on the Snellen chart at most recent exam

Exclusion Criteria:

1. Any central corneal pathology that could have impact on vision other than mild guttata felt unlikely to have any impact on corneal clarity.
2. Any documented glaucoma of any kind.
3. Any macular pathology except minimal drusen without retinal pigment epithelial pathology felt to be consistent with normal vision.
4. Any diabetic retinopathy other than minimal background diabetic retinopathy felt unlikely to affect vision.
5. Any other cause of central visual acuity loss including optic nerve, occipital cortex dysfunction or amblyopia.
6. Diagnosis of dry eye syndrome, defined as any corneal staining with fluorescein
7. Presence of any central posterior capsular opacification. Previous YAG laser capsulotomy is allowed.
8. Any surgical complication having to do with the capsule such as a broken capsule or zonular dialysis or iris trauma or any other complication felt to in any way impact upon the quality of the visual result.
9. Any contraindication to pupil dilation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Enrollment will be stratified into two patient groups based on time since surgery: (1) one to two years post-operative, and (2) two to three years post-op.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Light scattering | Post-opertative
  Correlation of random light scattering (measured with the C-Quant device) with severity of glistenings in the lenses

SECONDARY OUTCOMES:
Visual function | Post-operative
  Correlation of visual function (visual acuity, contrast acuity and constrast acuity with glare)with glistening severity
Visual quality | Post-operative
  Correlation of visual quality (measured with quality of life questionnaire, and subjective reports of symptoms) with glistening severity

CONTACTS AND LOCATIONS:
Overall Officials: Randall J Olson, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, John Moran Eye Center, Salt Lake City, Utah, United States